CLINICAL TRIAL: NCT04421352
Title: A Phase Ia/Ib, Open-Label, Multiple-Dose, Dose-Escalation and Expansion Study of the Anti-PD-L1 Monoclonal Antibody CS1001 in Subjects With Advanced Solid Tumors
Brief Title: Safety and Tolerability Evaluation of Low-dose Radiation in Combination With CS1001 in Relapsed SCLC Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1001-101-13
Record Dates: First submitted 2020-05-29; First posted 2020-06-09 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Relapsed Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- low-dose radiation+CS1001 (Experimental): low-dose radiation+CS1001
  Interventions: Drug: CS1001

INTERVENTIONS:
Drug: CS1001 — low-dose radiation+CS1001 1200mg Q3W. In the dose escalation part, the dose levels will be escalated following a modified 3+3 dose escalation scheme.
  Dose A: 3Gy/1f; Dose B: 9Gy/3f; Dose C: 15Gy/5f;
  In the dose expansion part, more SCLC patients will be assigned.

SUMMARY:
A Phase Ia/Ib Safety and Tolerability Evaluation of Low-dose Radiation in Combination with CS1001 in relapsed SCLC patients

DETAILED DESCRIPTION:
This is a dose-escalation study of Low-dose Radiation in combination with CS1001 in relapsed SCLC patients. Patients are assigned to 3 treatment groups received from 3 Gy to 15Gy, to determine the safety, tolerability and the maximal tolerant dose. Biomarkers and immunological markers are collected and analyzed as well.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed LS-SCLC or ES-SCLC and experienced progression since first-line standard platinum containing dual-drug chemotherapy.
2. Patients whose initial diagnosis was limited must undergo radical chest radiotherapy and the time of tumor progression is not less than 3 months from the end of radiotherapy, or cannot receive radical chest radiotherapy due to specific reasons
3. At least one extracranial measurable lesion (RECIST v1.1), and for a lesion that has received radiotherapy, progression of the lesion after radiotherapy must be confirmed.
4. Patients with brain metastases are allowed to receive previous radiotherapy and their condition is stable, but the time to the end of radiotherapy must not be less than 3 months.
5. No radiotherapy contraindications were judged by the radiologist
6. ECOG performance status of 0 or 1.
7. Patients with life expectancy ≥ 3 months.
8. Patients must have adequate organ function.
9. Fertile men and women of childbearing potential must agree to use an effective method of birth control from providing signed consent and for 6 months after last study drug administration.

Exclusion Criteria:

1. Subjects known to have primary CNS tumors or meningeal metastases or unstable CNS metastases.
2. Patients with active autoimmune diseases or history of autoimmune diseases should be excluded.
3. Patients who have received immune checkpoint proteins/antibody/medicine (including PD-1, PD-L1, etc) for treatment.
4. Known history of HIV infection.
5. Subjects with active chronic hepatitis B or active hepatitis C .
6. Patients who have serious hypersensitive reaction to monoclonal antibodies, and have history of uncontrolled allergic asthma.
7. Known history of alcoholism or drugs abuse.
8. Subjects with history of radiation pneumonitis of grade 3 or above, regardless of recovered or not.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
To determine the recommended radiation dose and preliminarily evaluate the anti-tumor efficacy of CS1001 in combination with low-dose radiotherapy in subjects with limited or extensive stage SCLC who failed the firstline treatment | From date of the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AE) and Dose-Limiting Toxicity (DLT) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) V4.03 | From first dose to 30 days after last dose of CS1001, up to 2 years.
Cmax: Peak concentration, the maximum drug concentration measured during one dosing cycle | From first dose to 30 days after last dose of CS1001, up to 2 years.
The number and percentage of subjects with detectable Anti-drug Antibody (ADA) | From first dose to 30 days after last dose of CS1001, up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Result] Horn L, Mansfield AS, Szczesna A, Havel L, Krzakowski M, Hochmair MJ, Huemer F, Losonczy G, Johnson ML, Nishio M, Reck M, Mok T, Lam S, Shames DS, Liu J, Ding B, Lopez-Chavez A, Kabbinavar F, Lin W, Sandler A, Liu SV; IMpower133 Study Group. First-Line Atezolizumab plus Chemotherapy in Extensive-Stage Small-Cell Lung Cancer. N Engl J Med. 2018 Dec 6;379(23):2220-2229. doi: 10.1056/NEJMoa1809064. Epub 2018 Sep 25. PMID 30280641
- [Result] Ready N, Farago AF, de Braud F, Atmaca A, Hellmann MD, Schneider JG, Spigel DR, Moreno V, Chau I, Hann CL, Eder JP, Steele NL, Pieters A, Fairchild J, Antonia SJ. Third-Line Nivolumab Monotherapy in Recurrent SCLC: CheckMate 032. J Thorac Oncol. 2019 Feb;14(2):237-244. doi: 10.1016/j.jtho.2018.10.003. Epub 2018 Oct 10. PMID 30316010
- [Result] Li LY, Wang H, Chen X, Li WQ, Cui JW. First-line atezolizumab plus chemotherapy in treatment of extensive small cell lung cancer: a cost-effectiveness analysis from China. Chin Med J (Engl). 2019 Dec 5;132(23):2790-2794. doi: 10.1097/CM9.0000000000000536. PMID 31856049
- [Result] Paz-Ares L, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Shire N, Jiang H, Goldman JW; CASPIAN investigators. Durvalumab plus platinum-etoposide versus platinum-etoposide in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): a randomised, controlled, open-label, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1929-1939. doi: 10.1016/S0140-6736(19)32222-6. Epub 2019 Oct 4. PMID 31590988
- [Result] Yin L, Xue J, Li R, Zhou L, Deng L, Chen L, Zhang Y, Li Y, Zhang X, Xiu W, Tong R, Gong Y, Huang M, Xu Y, Zhu J, Yu M, Li M, Lan J, Wang J, Mo X, Wei Y, Niedermann G, Lu Y. Effect of Low-Dose Radiation Therapy on Abscopal Responses to Hypofractionated Radiation Therapy and Anti-PD1 in Mice and Patients With Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2020 Sep 1;108(1):212-224. doi: 10.1016/j.ijrobp.2020.05.002. Epub 2020 May 15. PMID 32417411